CLINICAL TRIAL: NCT07231900
Title: Sodium Bicarbonate in Intra-dialytic Hypertension in Chronic Hemodialysis Patients
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Shani Zilberman Itskovich, Dr., Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0208-25-ASF
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hypertension in Dialysis Patients
Keywords: Intra-dialytic hypertension
MeSH Terms: interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium bicarbonate (Experimental): PO Sodium bicarbonate 500mg X2/day
  Interventions: Drug: Sodium Bicarbonate (NaHCO3)
- Placebo (Placebo Comparator): 1 tab X2/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Bicarbonate (NaHCO3) — Prescribing Sodium Bicaronate for intra-dualytic hypertension
  Arms: Sodium bicarbonate
Drug: Placebo — 1 tab X 2/day
  Arms: Placebo

SUMMARY:
The study is designed to diminish intra-dialytic hypertension in chrnic hemodialysis patients suffering from metabolic acidosis (low bicarbonate levels). The intervention is a tab of 500 mg sodium bicarbonate twice a day for one month, vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patient > 3 months
* 3 dialysis per week, KTV>1.2
* capable of informed concent.
* rise in blood pressure during hemodialysis > 10 mm Hg, for at least 50% of dialysis sessions in the month prior to inclusion.
* Normal volume status, by clinical physician assessment + bioimpedance

Exclusion Criteria:

* age under 18,
* pregnancy
* unable to sign informed concent
* planned for kidney transplant in the following 3 month.
* congestive heart failure (NYHA 3-4)
* hospitalization for acute MI or CHF in the past 3 months.
* low compliece to medical therapy
* regular pre-dialysis tests with bicarbonate > 24 in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 1 month
  Prevention of intra dialytic hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir medical center, Ẕerifin, Is, Israel

IPD SHARING:
Plan to Share IPD: Yes
blood pressure results, blood tests
Supporting Information: Study Protocol, SAP, CSR